CLINICAL TRIAL: NCT01037036
Title: An Open-Label, Phase 2 Study of the Latanoprost Punctal Plug Delivery System (L-PPDS) With Adjunctive Xalatan® Eye Drops in Subjects With Ocular Hypertension (OH) or Open-Angle Glaucoma (OAG)
Brief Title: A Study of the L-PPDS With Adjunctive Xalatan® Eye Drops in Subjects With OH or OAG
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mati Therapeutics Inc. (Industry)
Collaborators: QLT Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PPL GLAU 08
Record Dates: First submitted 2009-12-17; First posted 2009-12-21 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2013-12

CONDITIONS: Ocular Hypertension; Open-Angle Glaucoma
Keywords: Ocular Hypertension; Open-Angle Glaucoma; Xalatan; IOP
MeSH Terms: conditions — Ocular Hypertension; Glaucoma, Open-Angle | interventions — Latanoprost

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Latanoprost Punctal Plug Delivery System followed by Xalatan (Experimental): Subjects will have the Latanoprost Punctal Plug Delivery System placed for 4 week or until loss of efficacy. After removal of the Latanoprost Punctal Plug Delivery system, subjects will administer adjunctive Xalatan eye drops once daily for 2 weeks. This is a single arm study.
  Interventions: Drug: Latanoprost Punctal Plug Delivery System; Drug: Xalatan

INTERVENTIONS:
Drug: Latanoprost Punctal Plug Delivery System — To evaluate the control of IOP compared to baseline, for an experimental dose of Latanoprost Punctal Plug Delivery System for 4 week or until loss of efficacy. This is a single arm study.
Drug: Xalatan — Subjects will administer adjunctive Xalatan eye drops once daily for 2 weeks. This is a single arm study.

SUMMARY:
The objective of this study is to investigate how the intraocular pressure (IOP)-lowering effect of the L-PPDS is altered by adjunctive Xalatan therapy.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years
* Diagnosed with bilateral Open-Angle Glaucoma or Ocular Hypertension
* Currently on prostaglandin therapy

Exclusion Criteria:

* Uncontrolled medical conditions
* Subjects who wear contact lenses
* Subjects requiring chronic topical artificial tears, lubricants, and /or - requiring any other chronic topical medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-12; Primary Completion 2010-04 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in IOP measurements | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Cuzanni, MD, MSc, Study Director — QLT Inc.
Locations (1):
- Menlo Park, Menlo Park, California, United States